CLINICAL TRIAL: NCT05278884
Title: Can the VAST Course Enhance Resuscitation Skills in a Resource-limited Setting?
Brief Title: Can VAST Improve ACLS in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University of Rwanda (Other); ANZCA Health Equity Project (Unknown)
Responsible Party: Principal Investigator, Teresa Skelton, Anesthesiologist, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: TSkelton
Record Dates: First submitted 2022-02-28; First posted 2022-03-14 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Global Health; Education; Resuscitation

STUDY DESIGN:
Intervention Model Description: For each hospital, the intervention will be to pair a 2-day technical resuscitation skills training adapted from the ACLS/AHA and a 3-day VAST course for a multidisciplinary team of 20 participants (i.e., nurses, doctors, non-physician anesthesia providers). Participants' resuscitation skills will be tested at 4 time points: immediately before the ACLS course, immediately after the ACLS course, immediately after the VAST Course, and at 4 months post training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACLS and then VAST teaching intervention (Experimental): For each hospital, the intervention will be to pair a 2-day technical resuscitation skills training adapted from the ACLS/AHA and a 3-day VAST course for a multidisciplinary team of 20 participants (i.e., nurses, doctors, non-physician anesthesia providers). Participants' resuscitation skills will be tested at 4 time points: immediately before the ACLS course, immediately after the ACLS course, immediately after the VAST Course, and at 4 months post training.
  Interventions: Behavioral: Advanced Cardiac Life Support Training; Behavioral: Vital Anesthesia Simulation Training

INTERVENTIONS:
Behavioral: Advanced Cardiac Life Support Training — Advanced Cardiovascular Life Support (ACLS) is a resuscitation course to teach recognition and treatment of cardiopulmonary arrest in patients.
Behavioral: Vital Anesthesia Simulation Training — The Vital Anesthesia Simulation Training (VAST) Course focuses on core clinical practices and non-technical skills needed to respond to the most common urgent and emergent clinical challenges found in hospitals in resource-limited settings like Rwanda.

SUMMARY:
Aim The purpose of this study is to determine if the addition of the VAST Course to technical resuscitation skills training enhances healthcare providers' resuscitation performance in a resource-limited setting.

Objectives

The aims of this research will be achieved by meeting the following objectives:

1. Quantitative evaluation of study participants' resuscitation performance during a simulation scenario before ACLS course, immediately following ACLS course, immediately following VAST course, and at 4 months post training.
2. Qualitative exploration of the barriers and supports identified by course participants to implementing resuscitation in the workplace after resuscitation skills training through focus groups.

New knowledge Lessons learned from this study will help inform the design and the implementation of resuscitation training programs in resource-limited settings. This has potential to improve resuscitation capacity in resource-limited settings leading to higher quality of care for patients.

ELIGIBILITY:
Inclusion Criteria:

* Full course participation
* Available for focus group interviews

Exclusion Criteria:

* Refusal to provide informed consent
* Participated in VAST or ACLS training in the four months prior to study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Time to initiation of CPR | From start of simulation scenario to time of first chest compressions, assessment up to 2 minutes of simulation
  The time it takes for the team to start chest compressions in the simulation in seconds

SECONDARY OUTCOMES:
Time to epinephrine administration | From start of simulation scenario to time of first epinephrine administration, assessment up to 5 minutes of simulation
  The time it takes for the team to give epinephrine in the simulation in seconds
Time to defibrillation | From start of simulation scenario to time of first defibrillation, assessment up to 5 minutes of simulation
  The time it takes for the team to defibrillate in the simulation in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Skelton, MD, FRCPC, Principal Investigator — University of Toronto
Locations (1):
- University of Rwanda, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No
Final results will be prepared for publication but no plan to share IPD

REFERENCES:
- [Derived] Tuyishime E, Mossenson A, Livingston P, Irakoze A, Seneza C, Ndekezi JK, Skelton T. Resuscitation team training in Rwanda: A mixed method study exploring the combination of the VAST course with Advanced Cardiac Life Support training. Resusc Plus. 2023 Jun 16;15:100415. doi: 10.1016/j.resplu.2023.100415. eCollection 2023 Sep. PMID 37363124